CLINICAL TRIAL: NCT06149572
Title: Comparing Sitting Versus Lateral Position During Spinal Anesthesia Administration for Elective Cesarean Delivery on the Severity of Hypotension in Dessie Comprehensive Specialized Hospital, Ethiopia, 2023: a Randomized Controlled Trial
Brief Title: Comparing Sitting Versus Lateral Position During Spinal Anesthesia on the Severity of Hypotension:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Aynalem Befkadu Woldemichael, Woldemichael, Wollo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0778
Record Dates: First submitted 2023-09-28; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Severty of Hpotention
Keywords: Hypotention; Ethiopia; Dessie

STUDY DESIGN:
Intervention Model Description: the sitting and lateral groups followed and assessed parallelly
Who Masked: Investigator, Outcomes Assessor
Masking Description: The data collector and primary investigators will be blinded for the position of parturient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral (L) Position group (Experimental): Parturients will be put for spinal punctures at the lateral position
  Interventions: Procedure: lateral position procedure
- Sitting (S)position group (Active Comparator): Parturients will get spinal punctures at the Sitting position as comparison
  Interventions: Procedure: sitting position porocedure

INTERVENTIONS:
Procedure: lateral position procedure — Lateral positioning will be used as an intervention for spinal hypotension.
  Arms: Lateral (L) Position group
Procedure: sitting position porocedure — parturients will get spinal punctures in the sitting position
  Arms: Sitting (S)position group

SUMMARY:
This study aimed to assess the effect of sitting and lateral positions on the severity of hypotension during the initiation of spinal anesthesia in elective cesarean section. There will be Sitting and Lateral groups in the study.

DETAILED DESCRIPTION:
Source Population: All parturients who are scheduled for elective cesarean delivery under spinal anesthesia at Dessie Comprehensive Specialized Hospital

Sample size determination: This is the first study comparing siting and lateral positioning during the initiation of spinal anesthesia and no previous study was done in the study area. So the sample size is determined from a previous study done by Atashkhoei Simin et al.in Dubai in the same population with a reported incidence of hypotension of 50% in the lateral group and 76.6 % in a sitting position. Using G*Power (using version 3.1.9.2) with a power of 90%, confidence interval of 95%, and a ratio of treatment to control 1:1, it is estimated that 120 participants and considering dropping out and nonresponse (10% contingency) a total of 132 patients (66 in each group) would be needed. the investigators chose this paper because a large sample size was obtained using the G*Power application.

Sampling procedure A 7-month log book report showed 392 patients undergoing elective c/s. 120 patients will be recruited with a probability of 33% until the sample size is achieved by considering the sequential patients scheduled for C/S as the sampling frame. All patients have a 50% equal chance of being included in the study. The first patient will be recruited by lottery method and then every 3rd will be included until the required sample size is completed. After informed consent taken, eligible participants will be allocated to one of the two groups with a sealed non-transparent envelope containing the name of the study group.

Data collection procedures Three anesthetists will be trained by the principal investigator about how to collect the data for 10 days. The data collectors will explain the study and take written consent from each patient if they agree to participate in the study. Then the patient's fluid intake will be restricted and will run at 20ml/kg /hr.NS at the time of identification of cerebrospinal fluid as a co-loading via an 18-G intravenous Catheter. The study drug or placebo will be given 5 minutes before the spinal block. After applying the minimum standard monitoring like NIBP, ECG and pulse oximetry baseline HR and BP readings will be taken in the left lateral position, with the cuff positioned at the level of the heart. Then spinal anesthesia will be performed by a responsible anesthetist (who is blinded for the study) between L3-L4 interspace by using tuffurs line as a landmark with a 24 gauge spinal needle. After the free flow of cerebrospinal fluid (CSF), 12.5 mg of 0.5% isobaric bupivacaine (2.5 ml) and both groups of parturient will positioned supine with 15 degrees of left lateral tilt. Patients' socio-demographic data (age, sex, weight, BMI,), ASA, type of procedure, total amount of IV fluid, and duration of surgery will be recorded using a structured questionnaire. MAP and HR will recorded at 0 (baseline), 5, 10, 15, 20, 30, 40, 50, and 60 minutes intra-operatively in both exposed and unexposed groups. The requirement for vasopressors, antiemetic and anti-shivering like tramadol or pethidine will be studied during 15 intraoperative period and immediate postoperatively. Collected data will be checked for completeness, accuracy, and clarity by the principal investigator.

Blinding

The data collector and primary investigators will be blinded for the position of parturient.

The data collector will enter the OR after the spinal block is done. Random numbers which will be generated by computer software for all study participants will held in sealed envelopes until the day of surgery. On the day of surgery after they change clothes the mother will pick up the envelope that will opened by one anesthetist who will be responsible for writing the generated random number and letter as S for the Sitting group and L for the lateral position group by marker on the questioners.

Data quality management

Training will be given to data collectors regarding study tools, objectives of the study, rights of respondents, and confidentiality of the information. To ensure the quality of data, it will be checked out for completeness, accuracy, and clarity before data entry. The complete data will be entered into the SPSS version 22 computer program. Data clean-up and cross-checking will before analysis.

Data processing and statistical analysis

Data will be checked, coded, entered, and analyzed by SPSS version 22 computer program.

The normality of data will be checked by the Kolmogorov-Smirnov (K-S) test, histogram, Q-Q plot, box plot, kurtosis, and skewness. The presence of Outliers will also assessed by boxplot. Student t-test and Mann-Whitney test will be applied to compare continuous numerical variables of normally distributed and skewed data respectively. Statistical differences between groups for categorical data will analyzed using the Chi-squared test. Frequency, percentages, tables, and figures will be used to summarize data. Data will expressed in terms of mean ± SD for normally distributed data or median (inter quartile range) for skewed data. A P-value less than 0.05 is considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria

- American Society of Anesthesiologists Physical Status (ASA II)

Exclusion Criteria:

* Any contraindication for spinal anesthesia
* History of Hypertensive disorders, anemia, Heart disease, diabetes and placenta previa
* poly- or oligo-hydramnios
* Obesity (BMI ≥29-35 kg/m2)
* Height <155 cm
* multiple pregnancy
* Sample size and sampling procedure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 132 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Effect of Positioning on the Severity of Spinal-Induced Hypotension | Each participant will be followed 4 weeks
  severity of hypotension will be measured by blood pressure as it defined milled hypotension when mean arterial pressure is 20% below the baseline, moderate hypotension when below 20% to 30% and Severe hypotension is a decrease of mean arterial pressure greater than 30% below the Baseline

SECONDARY OUTCOMES:
Consumption of vasopressor. | Each participant will be followed a minimun of 4 weeks
  Consumption of vasopressor measured in mg/kg.
Grade of motor blockage: | Each participant will be followed 4 weeks
  Motor blockage grade will be measured according to the Bromage score which ranks from grade one to four.
level of sensory block: | Each participant will be followed 4 weeks
  level of block is measyloss of sharp sensation to pinprick bilaterally at the mid axillary

CONTACTS AND LOCATIONS:
Overall Officials: Aynalem Woldemichael, MSC, Principal Investigator — Wollo Universty
Locations (1):
- Dessie comprehensive specilized hospital, Dessie, Amhara, Ethiopia